CLINICAL TRIAL: NCT02352870
Title: Intervention for Improving Psychological Distress in Dialysis (iDiD) Feasibility Two Arm Randomised Controlled Trial: Online Cognitive Behavioural Therapy (CBT) Intervention With Therapist Support vs Online CBT Intervention Alone (no Therapist Support)
Brief Title: Intervention for Improving Psychological Distress in Dialysis
Acronym: iDiD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: National Health Service, United Kingdom (Other Government); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PAHTMZA WPAH 68913; 14.LO.1934 (Other: NHS research ethics committee)
Record Dates: First submitted 2015-01-22; First posted 2015-02-02 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2015-09

CONDITIONS: Kidney Failure, Chronic; Depression; Anxiety
Keywords: Feasibility study; Randomised controlled trial; Cognitive behavioural therapy; Psychological distress; Cognitive illness representations; Common sense model
MeSH Terms: conditions — Kidney Failure, Chronic; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerised CBT with therapist support (Experimental): Participants complete seven online cognitive behavioural therapy sessions weekly plus they receive three telephone support calls. The content of each of the sessions are summarised below:
  Session 1: Psycho-education about end-stage renal failure Session 2: Generation of CBT "hot cross bun" model of psychological distress Session 3: Coping strategies for managing negative emotions, including: acceptance, relaxation, expression and tips for improving sleep quality.
  Session 4: Identifying and challenging unhelpful thoughts Session 5: Goal setting and problem solving Session 6: Managing difficult social relationships Session 7: Progress recap and preparing for the future
  In addition to completing the seven online sessions the intervention arm received three 30 minute telephone support calls at weeks two, four, and six to facilitate engagement and understanding of the contents of the website.
  Interventions: Behavioral: Computerised Cognitive Behavioural Therapy; Behavioral: Telephone support
- Computerised CBT without therapist support (Active Comparator): Participants complete seven online cognitive behavioural therapy sessions weekly but do not receive any telephone support calls. The content of each of the sessions are summarised below:
  Session 1: Psycho-education about end-stage renal failure Session 2: Generation of CBT "hot cross bun" model of psychological distress Session 3: Coping strategies for managing negative emotions, including: acceptance, relaxation, expression and tips for improving sleep quality.
  Session 4: Identifying and challenging unhelpful thoughts Session 5: Goal setting and problem solving Session 6: Managing difficult social relationships Session 7: Progress recap and preparing for the future
  Interventions: Behavioral: Computerised Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Computerised Cognitive Behavioural Therapy — Online treatment sessions are scheduled to last approximately one hour, completed independently by the participant on a weekly basis
Behavioral: Telephone support — Telephone support calls are scheduled to last 30 minutes and and are received fortnightly at weeks: 2, 4 and 6.
  Arms: Computerised CBT with therapist support

SUMMARY:
To explore whether it is feasible to recruit and retain haemodialysis patients into a randomised controlled trial of online cognitive-behavioural therapy to manage distress

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over and receive hospital haemodialysis three-times weekly
2. Presence of mild to moderately severe depressive symptoms (based on PHQ-9 scores of 5 to 19 in range; a self-report measure of depression) and/or presence of mild to moderate anxiety symptoms (based on GAD-7 scores of 5-14)
3. Speak English sufficiently well to engage with screening tools
4. Have a basic understanding of how to use the Internet and an email address
5. Have a minimum dialysis vintage of ≥3 months (electronic patient record)

Exclusion Criteria:

1. Hospitalised at the time of assessment or within 1 month prior to the assessment
2. Currently receiving active treatment for depression and/or anxiety. We consider active treatment to be any current psychological treatments (talking therapies) or receipt of a new anti-depressant and/or anti-anxiety medication. A medication is considered new if it is commenced three months prior to the completion of the depression and anxiety screening questionnaire
3. Severe mental health disorders, for example, psychosis, bi-polar disorder
4. Active suicidal thoughts-any participant that scores greater than one on the depression PHQ-9 item "Thoughts that you would be better off dead, or of hurting yourself" will be excluded from the study.
5. Evidence of addiction to alcohol or drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Consent to psychological screen rate using self-report measures of depression (PHQ-9) and anxiety (GAD-7) | Baseline recruitment/screening
  Record the number of patients approached for screening and their consent rate

SECONDARY OUTCOMES:
Recruitment , randomisation, and retention rates | Screening, baseline, and 12 weeks follow-up
  Descriptive statistics as per CONSORT flow diagram
Adherence to the online intervention + telephone support calls (therapist supported arm only) | 12 weeks follow-up
  Number of online sessions accessed and their duration + number of calls completed and their duration (therapist supported arm only)
PHQ-9 (A self-report 9 item measure of depression) | Change in depression from baseline to 12 weeks
  A self-report 9 item measure of depression
GAD-7 (A self-report 7 item measure of anxiety) | Change in anxiety from baseline to 12 weeks
  A self-report 7 item measure of anxiety
EQ-5D (A self-report measure of quality of life) | Baseline and 12 weeks follow-up
  A self-report measure of quality of life
Brief Illness Perceptions Questionnaire | Baseline and 12 weeks follow-up
  A self-report measure of beliefs about illness
Client Service Receipt Inventory (A self-report measure of health service utilisation) | Baseline and 12 weeks follow-up
  A self-report measure of health service utilisation
Satisfaction with treatment (A 2 item measure generated for the purposes of present study) | Baseline and 12 weeks follow-up
  A 2 item measure generated for the purposes of present study

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chilcot, PhD, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Hudson JL, Moss-Morris R, Game D, Carroll A, Chilcot J. Improving Distress in Dialysis (iDiD): A tailored CBT self-management treatment for patients undergoing dialysis. J Ren Care. 2016 Dec;42(4):223-238. doi: 10.1111/jorc.12168. Epub 2016 Jul 26. PMID 27458126
- [Derived] Hudson JL, Moss-Morris R, Norton S, Picariello F, Game D, Carroll A, Spencer J, McCrone P, Hotopf M, Yardley L, Chilcot J. Tailored online cognitive behavioural therapy with or without therapist support calls to target psychological distress in adults receiving haemodialysis: A feasibility randomised controlled trial. J Psychosom Res. 2017 Nov;102:61-70. doi: 10.1016/j.jpsychores.2017.09.009. Epub 2017 Sep 21. PMID 28992899
- [Derived] Chilcot J, Hudson JL, Moss-Morris R, Carroll A, Game D, Simpson A, Hotopf M. Screening for psychological distress using the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS): Initial validation of structural validity in dialysis patients. Gen Hosp Psychiatry. 2018 Jan-Feb;50:15-19. doi: 10.1016/j.genhosppsych.2017.09.007. Epub 2017 Sep 28. PMID 28985589